CLINICAL TRIAL: NCT04138030
Title: Conventional Versus Cold Snare Endoscopic Mucosal Resection of Colonic Lateral Spreading Lesions - A Randomised Controlled Trial
Brief Title: Conventional Endoscopic Mucosal Resection Versus Cold Snare Endoscopic Mucosal Resection of Colonic Lateral Spreading Lesions - A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Professor, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (6114) 2019/ETH11826
Record Dates: First submitted 2019-10-20; First posted 2019-10-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Adenoma Colon; Colon Adenoma; Colon Cancer
Keywords: Colonoscopy; Polypectomy; Adenoma; Colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Adenoma; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Endoscopic Mucosal Resection (Active Comparator): Conventional Endoscopic Mucosal Resection (EMR), if necessary, to 15-40mm laterally spreading adenomas.
  Interventions: Procedure: Conventional Endoscopic Mucosal Resection
- Cold Snare Endoscopic Mucosal Resection (Active Comparator): Cold Snare Endoscopic Mucosal Resection (EMR), if necessary, to 15-40mm laterally spreading adenomas.
  Interventions: Procedure: Cold Snare Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Conventional Endoscopic Mucosal Resection — Use of injected chromogelofusine solution to raise a lesion prior to polypectomy snare closed over a polyp with electrocautery
  Other Names: Conventional EMR
  Arms: Conventional Endoscopic Mucosal Resection
Procedure: Cold Snare Endoscopic Mucosal Resection — Use of injected chromogelofusine solution to raise a lesion prior to polypectomy snare closed over a polyp without electrocautery
  Other Names: CSP
  Arms: Cold Snare Endoscopic Mucosal Resection

SUMMARY:
Comparing the complete resection rate and subsequent adenoma recurrence rate at surveillance colonoscopy of 15-40mm laterally spreading adenomas for conventional EMR vs. cold snare EMR.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common malignancy worldwide and the fourth leading cause of cancer related death, with rates being highest in Western countries. Colonoscopy is considered the golden standard in colorectal cancer screening and endoscopic resection of precursor lesions (polyps) has been shown to reduce colorectal cancer death. Polyps extending over 10mm, also referred to as lateral spreading lesions (LSL) if non-pedunculated, more often demonstrate advanced histological features and are considered to be at greater risk for malignant transition as compared to their smaller counterparts. Incomplete endoscopic resection of advanced adenomas may lead to adenoma recurrence and contribute to the development of so called 'interval cancers', which occur during the 6 - 36 month period following complete colonoscopy. Interval cancers account for up to 6% of newly diagnosed CRC cases, highlighting the importance of complete resection.

Endoscopic mucosal resection (EMR) is a well-established inject and resect method for the removal of LSLs using chromo-gelofusin based submucosal lift and subsequent cauterisation assisted snare excision. Lesions up to 25mm in size may be removed enbloc, whereas larger lesions are generally removed in a piecemeal fashion. Contrary to enbloc resection, piecemeal EMR is historically associated with relatively high recurrence rates of 15-20%. A recent four centre trial led by Westmead Hospital published in gastroenterology (impact factor 20.8) has shown that application of snare-tip soft coag (STSC) to the EMR defect margins considerably improves recurrence rates to around 7% in adenomatous LSL. Common complications of EMR such as intra-procedural bleeding (IPB) or clinically significant post-procedural bleeding (CSPB), deep mural injury (DMI) and post-polypectomy coagulation syndrome (PPCS) are largely related to the use of cauterisation for tissue transection. Although complication rates have improved and effects can often be managed endoscopically, further optimization of the EMR safety profile is needed in the background of an aging target population with multiple co-morbidities and widespread use of anticoagulants.

Cold snare polypectomy (CSP) has become the standard of care for removal of subcentimeter polyps. CSP relies on the use of dedicated stiff thin wire snares that are able to swiftly cut through mucosal tissue without the need for cauterisation, leaving intact the muscularis mucosa and the deeper submucosal layers, virtually excluding the risk of perforation. The absence of delayed cauterisation effect significantly reduces the risk of post-polypectomy bleeding, even in patients on anticoagulant therapy. Complete resection rates of polyps ranging from 6 to 10mm in size were found to be non-inferior in CSP as compared to cauterisation based resection. Moreover, resecting a sufficient margin of normal mucosa surrounding the polyp (i.e. >1mm) yields an excellent 98% complete resection rate in polyps <10mm in size without increasing the risk of delayed bleeding. Meta-analysis demonstrated a significantly shorter procedure time when applying the cold snare resection technique in small polyps. Snare size limitations of dedicated cold snares however do not allow for en-bloc resection of polyps >10mm.

Recently, cold snare piecemeal EMR was shown to be safe and effective for the removal of large sessile serrated polyps (SSP). Combined evidence from a limited number of small single centre mostly retrospective studies investigating cold snare piecemeal polypectomy in adenomas over 10mm demonstrated recurrence rates of around 11% whilst maintaining an excellent safety profile with minimal complication rates. However, recurrence rates rise to 22% in the subgroup of polyps over 20mm. Thus far cold snare piecemeal polypectomy of lateral-spreading adenomas has not yet been compared to conventional EMR in prospective randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing colonoscopy who is older than 18 years of age, has a written consent for trial participation and has at least one LSL meeting to the following description:

  * Localisation in the colon or rectum
  * Benign adenomatous surface features (Kudo III / IV, JNET 2a)
  * Granular or non-granular topography
  * Paris classification 0-IIa/IIb +/- Is
  * If present, sessile component may be no greater than 10mm in size.
  * Polyp size ranging from 15 to 40mm

Exclusion Criteria:

* Current use of antiplatelet (excluding aspirin) or anticoagulants which have not appropriately been interrupted according to the guidelines.
* Known bleeding disorder or coagulopathy.
* Pregnancy
* History of inflammatory bowel disease
* Previously attempted or otherwise non-lifting lesions
* Endoscopic features suggestive of submucosal invasion (Kudo Vi/n, JNET 2b / 3) or concurrent CRC
* Lesions involving the ileocaecal valve (ICV) or the anorectal junction (ARJ)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Complete resection rate | 1 day
  Complete resection rate (CRR) as determined by endoscopic assessment (no visible residual adenoma) and histological assessment (biopsies of resection margin)
Adenoma recurrence rate | 4-6 months
  Adenoma recurrence rate (ARR) at SC1 as determined by endoscopic assessment (no visible recurrent adenoma) and histological assessment (scar biopsies)

SECONDARY OUTCOMES:
Time to perform polypectomy | 1 day
  Time needed to perform polyp resection measured from first snare positioning until complete resection is achieved based on endoscopic assessment, and total procedure time from insertion of the scope until all specimens have been collected and the scope withdrawal is completed.
Intra-procedural and post-procedural complications | 30 days
  Intra-procedural and post-procedural complications rates (IPB / CSPB / DMI / PPCS) as previously described

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, Principal Investigator — Western SLHD
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] O'Sullivan T, Cronin O, van Hattem WA, Mandarino FV, Gauci JL, Kerrison C, Whitfield A, Gupta S, Lee E, Williams SJ, Burgess N, Bourke MJ. Cold versus hot snare endoscopic mucosal resection for large (>/=15 mm) flat non-pedunculated colorectal polyps: a randomised controlled trial. Gut. 2024 Oct 7;73(11):1823-1830. doi: 10.1136/gutjnl-2024-332807. PMID 38964854